CLINICAL TRIAL: NCT03177291
Title: A Phase I/Ib Trial of Pirfenidone Combined With Standard First-Line Chemotherapy in Advanced-Stage Lung NSCLC
Brief Title: Pirfenidone Combined With Standard First-Line Chemotherapy in Advanced-Stage Lung NSCLC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-19082
Record Dates: First submitted 2017-06-02; First posted 2017-06-06 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Lung Cancer; Non Small Cell Lung Cancer; Advanced Cancer; Metastatic Lung Cancer; Squamous Cell Lung Cancer; Non-Squamous Non-Small Cell Neoplasm of Lung
Keywords: NSCLC; SCLC
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — pirfenidone; Carboplatin; Paclitaxel; Albumin-Bound Paclitaxel; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Squamous Cell Lung Cancer (SQCLC) (Active Comparator): Arm A Combination Therapy: Pirfenidone combined with standard first-line chemotherapy. Participants will receive the combination of Pirfenidone and carboplatin plus paclitaxel in study treatment cycles that last 21 days. Phase 1 Dose Escalation; followed by Phase 1b Dose Expansion.
  Interventions: Drug: Pirfenidone; Drug: Carboplatin; Drug: Paclitaxel
- Non-Squamous Cell Lung Cancer (SQCLC) (Active Comparator): Arm B Combination Therapy: Pirfenidone combined with standard first-line chemotherapy. Participants will receive the combination of Pirfenidone and carboplatin plus pemetrexed in study treatment cycles that last 21 days. Phase 1 Dose Escalation; followed by Phase 1b Dose Expansion.
  Interventions: Drug: Pirfenidone; Drug: Carboplatin; Drug: Pemetrexed

INTERVENTIONS:
Drug: Pirfenidone — Pirfenidone: 267 mg Capsules by mouth (PO) 3 times per day (TID). Dose Escalation: Level 1:One capsule (total daily dose 801 mg); Level 2: Two capsules (total daily dose 1602 mg); Level 3: Three capsules (total daily dose 2403 mg).
  Dose Expansion: Treatment at dose determined by the Phase 1 Dose Escalation.
  Other Names: 5-methyl-1-phenyl-1H-pyridine-one; Esbriet
Drug: Carboplatin — Area under the curve (AUC) 6 on Day 1 of a 21-day cycle for 4 - 6 cycles.
  Other Names: Paraplatin
Drug: Paclitaxel — 200 mg/m^2 on Day 1 of a 21-day cycle for 4 - 6 cycles.
  Other Names: Abraxane
  Arms: Squamous Cell Lung Cancer (SQCLC)
Drug: Pemetrexed — 500 mg/m^2 on Day 1 of a 21-day cycle for 4 - 6 cycles.
  Other Names: Alimta
  Arms: Non-Squamous Cell Lung Cancer (SQCLC)

SUMMARY:
The purpose of this study is to find out what effects (good and/or bad) Pirfenidone combined with standard first-line chemotherapy will have on you and non-small cell lung cancer (NSCLC). The investigational drug Pirfenidone is being combined with standard chemotherapy in participants with advanced non-small cell lung cancer. Pirfenidone is approved to treat idiopathic pulmonary fibrosis (IPF) but it isn't currently approved to treat non-small cell lung cancer.

DETAILED DESCRIPTION:
This study will be conducted in two phases: 1) a Phase I dose escalation study with a Standard 3+3 design to determine the recommended Phase II dose and 2) a Phase Ib expansion study to evaluate early signs of efficacy and obtain more toxicity data. The Phase I trial will be a single center, dose-escalation study of pirfenidone combined with standard chemotherapy in the treatment of advanced/metastatic NSCLC, followed by a Phase Ib trial to determine early clinical efficacy [objective tumor response rate (ORR)] and toxicity data.

ELIGIBILITY:
Inclusion Criteria:

* Histologically/cytologically documented Stage IIIB to Stage IV unresectable non-small cell lung cancer (either squamous cell carcinoma or non-squamous cell lung cancer or mixed histology; epidermal growth factor (EGFR) or ALK mutation excluded unless previously treated with a TKI, given a 2 week washout period). Patients with adenocarcinoma must have been tested for EGFR and ALK mutations.
* At least one measurable tumor lesion as defined by Response Evaluation Criteria In Solid Tumors (RECIST) v1.1.
* 18 years of age and older.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Participants should be chemotherapy naïve in the Stage IV NSCLC setting, with the exception of chemotherapy for neoadjuvant or adjuvant treatment that completed at least 6 months before the study treatment.
* Participants' blood test must meet the following requirements: Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L; Platelets ≥ 100 x 10^9/L; Hemoglobin level ≥ 9 g/dL.
* Clinical biochemistry examination must meet the following requirements: Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x upper limit of normal (ULN) or ≤ 5 X ULN for patients with liver metastases; Serum creatinine ≤ 1.5 x ULN or estimated GFR ≥ 50 mL/min/m^2; Total bilirubin ≤ 1.5 x ULN; Urine pregnancy test is negative for women of childbearing potential, within 14 days before study treatment.
* Estimated life expectancy of at least 6 months.
* May have received prior immunotherapy.
* Have archived tissue available or be willing to undergo a fresh biopsy during screening, if deemed feasible by the investigator/study PI. If neither available, the patients enrollment must be reviewed and approved by the PI.
* Voluntarily participate in the clinical trial, understanding they may withdraw participation at any time.
* Able to understand and provide written informed consent prior to trial participation.

Exclusion Criteria:

* Are currently undergoing other anti-tumor therapies or have concurrent active cancer.
* Patients who were enrolled into any other treatment clinical trial and received treatment on that trial within 4 weeks of study treatment.
* Any clinical laboratory findings give reasonable suspicion of a disease or condition that contraindicates the use of any study medication or render the subject at high risk from treatment.
* Patients with previously untreated brain metastases should be excluded. Patients with treated and stable (>4 weeks) brain metastases may be eligible for enrollment.
* History of allergic reactions to carboplatin or paclitaxel.
* Have had immunotherapy or radiotherapy within 4 weeks prior to study treatment or those who have not recovered from adverse events due to agents administered more than 4 weeks prior to study treatment. Prior history of palliative radiation for symptomatic bony or brain metastases is permissible.
* Are receiving any other investigational agents.
* Patients with known ROS1 mutations who have not received prior targeted therapy.
* Alcohol or drug dependence.
* Uncontrolled coagulopathy.
* Uncontrolled hyper- or hypothyroidism.
* Known hypersensitivity to pirfenidone, carboplatin, pemetrexed or paclitaxel.
* Pre-existing peripheral neuropathy of Grade II or higher.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure (NYHA Class III/IV), unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients receiving any medications or substances that are moderate to strong inhibitors CYP1A2 are ineligible.
* Pregnant women are excluded from this study. Women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of study drug administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-09-26 (Actual); Primary Completion 2021-05-09 (Actual); Study Completion 2024-12-04 (Actual)

PRIMARY OUTCOMES:
Phase 1: Recommended Phase 1b Dose | 6 months post final enrollment in phase 1 - up to 48 months
  Recommended Phase 1b dose of Pirfenidone in combination with standard first-line chemotherapy, based on Dose Limiting Toxicity (DLT) from phase 1. Dose-limiting Toxicity: The occurrence of any of the following toxicities will be considered a DLT, if judged by the Investigator to be possibly, probably, or definitely related to study drug administration, referring to grade 3-5 adverse events as listed in the protocol document.
Phase 1b: Overall Response Rate (ORR) | 6 months post final enrollment in phase 1b - up to 48 months
  ORR according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1: Complete Response (CR) plus Partial Response (PR). Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm (<1 cm). Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Up to 48 months
  PFS according to RECIST 1.1: defined as the time from study registration to progression or death, whichever comes first. PFS for patients last known to be alive and progression free will be censored at the date of last disease assessment. Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm (0.5 cm).
  (Note: the appearance of one or more new lesions is also considered progressions). Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Overall Survival (OS) | Up to 48 months
  Overall survival (OS) defined as the time from study registration or death due to any cause. OS for patients last known to be alive will be censored at the date of last contact.

CONTACTS AND LOCATIONS:
Overall Officials: Jhanelle Gray, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials website — https://moffitt.org/clinical-trials-research/